CLINICAL TRIAL: NCT05206188
Title: Mastering the World of Work (MWW): Randomized Controlled Trial
Brief Title: Mastering the World of Work (MWW): RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6377E
Record Dates: First submitted 2021-12-14; First posted 2022-01-25 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Mental Disorders; Employment; Metacognition; Employment, Supported
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Study participants randomized to the experimental condition will receive IPS services in combination with the MWW intervention. Study participants randomized to the control condition will receive IPS services as usual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Study participants randomized to the experimental condition will receive IPS services as usual in conjunction with the MWW intervention.
  Interventions: Behavioral: Mastering the World of Work (MWW)
- Control (No Intervention): Study participants randomized to the control condition will receive IPS services as usual.

INTERVENTIONS:
Behavioral: Mastering the World of Work (MWW) — Mastering the World of Work (MWW) is a 29-session individual intervention comprised of 7 modules each covered in 4 sessions, and a wrap-up session. Participants in the randomized clinical trial will be offered to meet on a weekly basis with the MWW clinician assigned to work with them.
  Arms: Experimental

SUMMARY:
The purpose of this study is to conduct a randomized clinical trial for an innovative intervention entitled "Mastering the World of Work" (MWW). MWW aims to improve the employment outcomes of individuals with psychiatric disabilities who experience metacognitive deficits. Metacognitive deficits are represented in diminished capacity to form an integrated sense of self and others and respond to challenges in life. The randomized trial (N=60) will be conducted with recipients of Supported Employment (Individual Placement and Support) services at the Mental Health Center of Greater Manchester, in Manchester, NH. Given COVID-19 safety considerations, the MWW intervention will be delivered in a hybrid manner depending on the preferences of both clinicians and clients at the MHCGM at any given point of the study. The feasibility of remote delivery of the intervention has been established as part of a pilot study conducted at BU CPR. Thus, clinicians may deliver the intervention using HIPAA-complaint ZOOM connection and/or in person. The assessments will be administered at baseline, 6, 12, and 18 months post baseline remotely by BU staff using a HIPAA-complaint ZOOM connection. The RCT will establish preliminary evidence about the incremental effectiveness of the MWW intervention to improve the employment outcomes of individuals with metacognitive deficits who receive high fidelity IPS services. Study participants randomized to the control condition will receive IPS services as usual.

DETAILED DESCRIPTION:
Mastering the World of Work (MWW) is a 29-session individual intervention comprised of 7 modules each covered in 4 sessions, and a wrap-up session. The 7 modules address: i) awareness of one's motivations to work; ii) awareness about personal work-related strengths and vulnerabilities; iii) balancing between work and mental health; iv) understanding experience of workplace prejudice and discrimination; v) understanding work-related challenges such as workload, time management, etc.; vi) understanding conflicts at work; and vii) thoughts and feelings about receiving disability benefits and their impact on work-related decisions. The last module is optional for individuals who receive disability benefits due to their psychiatric condition. Each session includes viewing a short video depicting the session's concept followed by a discussion of how it is applicable to the participant's life. Sessions can last up to one hour depending on participant's speed of covering the session's material. Findings from the feasibility study indicate that on average MWW sessions last between 30 and 45 minutes. Participants will complete a homework assignment related to each topic discussed in-between sessions; this will take participants an average of 15-20 minutes per week.

Participants in the randomized clinical trial will be offered to meet on a weekly basis with the MWW clinician assigned to work with them. Participants can choose to have the MWW sessions delivered remotely or in person in a flexible manner that fits the preferences and safety concerns of both the client and the clinician at any given point of the study. Participants will be able to meet in person at the MHCGM agency or remotely via a HIPAA-compliant Zoom connection. Participants will be reminded that MWW sessions will be audio-recorded and audio files will be shared with the BU research team for the purposes of supervision and fidelity assessment as indicated in the consent form the participants have signed.

The MWW intervention will be delivered in a flexible manner informed by the feasibility study conducted at BU CPR which demonstrated that it is important to schedule sessions depending on participants' personal situation and preferences. Occasionally, participants may need two meetings to cover the content of a given session or alternatively, may cover in one meeting the content of two sessions within a given module if the content is not particularly relevant to their personal situation (i.e., the participant reports not having experiences of prejudice and discrimination at work). Participants will be able to cover MWW modules out of order depending on their employment situation, i.e., a participant may choose to complete the module on conflict at work (module 6) earlier if that participant gets a job and right away encounters a conflict with a co-worker or a supervisor. Participants may reschedule meetings due to any personal/medical reasons or take a break due to changes in their employment situation (i.e., getting a full-time job). Clinicians will be available to meet with participants during all 18 months of their study participation. Once participants complete all relevant MWW modules, participants can still continue to meet with their clinician to go over some MWW content relevant to the participant's employment situation. Participants can schedule such follow-up sessions as frequently as necessary while accounting for their clinician's availability at the time of such requests.

Each participant will be in the study for 18 months and will complete a total of 4 assessments over the course of the study: at baseline, 6-month, 12-month and 18-month post-baseline. The baseline assessment will last approximately between 90 minutes and 2 hours and the follow-up assessments will take approximately 60 to 90 minutes.

The MWW intervention sessions will also be audio recorded. BU Research Staff will review a percentage of these recordings to assess fidelity, that is, to ensure that key components of the session were covered. The BU Research Staff will also review these recordings for the supervision of the clinicians delivering the MWW intervention.

ELIGIBILITY:
Inclusion Criteria:

1. are 18 or older
2. have a DSM-IV diagnosis of serious mental illness, including dual diagnosis
3. are currently receiving supported employment services (Individual Placement and Support) at the Mental Health Center of Greater Manchester, in Manchester, NH.
4. are not currently employed for one of the following three reasons: i. newly enrolled in IPS and have not yet been placed in a job ii. have been enrolled in IPS for at least three months and have not yet obtained a job iii. have lost a job after enrollment in IPS and have not obtained a new job for at least a month following the loss of their last job.
5. are fluent in English
6. are able and willing to participate via Zoom in assessments and if necessary in intervention delivery
7. agree that assessments and intervention sessions will be audio-recorded

Exclusion Criteria:

1. inability to give full and knowing consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-24 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Employment Rates | 18 months
  Obtainment of a competitive job
Employment Tenure | 18 months
  Number of weeks during which participant kept a job: remained on payroll either due to earned income (at least 1 hour of paid work) or used vacation and/or sick time.

SECONDARY OUTCOMES:
Metacognition Assessment Scale - Abbreviated (MAS-A) | 18 months
  Metacognition Assessment Scale - Abbreviated (MAS-A) is a rating scale measuring metacognitive capacity with 4 subscales assessing: a) self-reflectivity; b) awareness of the other's mind; c) decentration; and d) mastery. The scores for the overall MAS-A scale range between 0 and 28 with higher scores indicating higher level of metacognitive capacity. The scores for the MAS-A subscales range as follows with higher scores indicating higher level of specific metacognitive capacity: a) self-reflectivity - between 0 and 9; b) awareness of the other's mind - between 0 and 7; c) decentration - between 0 and 3; and d) mastery - between 0 and 9.

CONTACTS AND LOCATIONS:
Overall Officials: Zlatka Russinova, PhD, Principal Investigator — Boston University Center for Psychiatric Rehabilitation
Locations (1):
- Mental Health Center of Greater Manchester, Manchester, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Yes
We will follow the guidance outlined in the Administration for Community Living (ACL) Public Access Plan for peer-reviewed publications and establishing public access to data. We will use the Interuniversity Consortium for Political and Social Research (ICPSR) as designated by ACL for archiving of data.
Time Frame: Data will be shared upon study completion without availability limits.
Access Criteria: Not available yet.